CLINICAL TRIAL: NCT06971445
Title: Effect of Polyunsaturated Fatty Acids Omega-3 Supplementation on Pregnancy Outcomes and Inflammation Markers in Pregnant Women HIV+, With Antiretroviral Therapy, Randomized Clinical Trial.
Brief Title: Effect of Omega-3 Supplementation on Pregnant Outcomes and Inflammation Markers of Women Infected With HIV Using Antiretroviral Therapy
Acronym: OM3HIVPROUTINF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, Estela Ytelina Godínez Martínez, Researcher in Medical Science B, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-1-40; 2024-1-40 (Other: Instituto Nacional de Perinatologia)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pregnant HIV Positive Women
Keywords: Dietary Supplements; Fatty Acids, Omega-3; pregnancy outcomes; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 polyunsaturated fatty acids (PUFA n-3) (Experimental): 1280 mg Polyunsaturated Fatty Acid n3 (650mg EPA, 450mg DHA and179mg ALA) per day for 8 weeks
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids (PUFA n-3)
- Olive oil (Active Comparator): Olive oil softgels with a similar appearance to the experimental softgels (PUFA n-3) for 8 weeks
  Interventions: Dietary Supplement: Olive oil (placebo)

INTERVENTIONS:
Dietary Supplement: omega-3 polyunsaturated fatty acids (PUFA n-3) — 1280 mg of omega-3 polyunsaturated fatty acids (650mg EPA, 450mg DHA, and 179mg ALA) per day for 8 weeks
  Arms: omega-3 polyunsaturated fatty acids (PUFA n-3)
Dietary Supplement: Olive oil (placebo) — Softgels containing extra virgin olive oil, with a similar appearance to the experimental group, were given to participants for 8 weeks.
  Arms: Olive oil

SUMMARY:
This clinical trial aims to determine the effect of PUFA-n3 supplementation on birth weight, gestational length, and plasma inflammatory markers in pregnant women with HIV who are on antiretroviral therapy. The key questions this study seeks to answer are:

1. Will the neonates of HIV-positive women who received 1280 mg of PUFA-n3 supplementation during pregnancy have higher birth weights and longer gestation periods compared to the neonates of HIV-positive women who received a placebo?
2. Will the inflammatory markers in HIV-positive women who received 1280 mg of PUFA-n3 during pregnancy differ from those of HIV-positive women who received a placebo?

Researchers will compare the effects of 1280 mg of PUFA-n3 supplementation against a placebo (olive oil) to determine if the supplement can increase birth weight, gestational length, and attenuate the inflammation.

Participants in the study will:

* Take a prenatal multivitamin that includes 300 mg of PUFA-n3
* Take either 1280 mg of PUFA-n3 or a placebo daily for 8 weeks, starting from a gestational age of 20-29 weeks.
* Visit the hospital at the beginning of the study and again 8 weeks later for blood sampling. Additionally, they will have follow-up visits every 2 weeks to monitor gestational weight gain and dietary intake.
* Keep a diary to register their supplement intake and record any side effects.

DETAILED DESCRIPTION:
In pregnant women infected with human immunodeficiency virus (HIV), antiretroviral therapy (ART) during pregnancy significantly reduces the risk of neonatal or vertical transmission of the virus. However, these women may face a higher risk of adverse outcomes for their babies, including preterm birth, low birth weight, and being small for their gestational age. HIV infection and ART contribute to a chronic inflammatory state, which has been linked to these negative pregnancy outcomes.

Additionally, the typical diet of pregnant women receiving perinatal care at the Instituto Nacional de Perinatología often lacks sufficient polyunsaturated fats. This is primarily due to limited access to a diverse and high-quality diet, which is frequently influenced by their socioeconomic status. Supplementation with polyunsaturated omega-3 fatty acids (PUFA-n3) during pregnancy has been proposed as a preventive measure against adverse outcomes such as preterm birth and low birth weight. Several studies have documented the efficacy of PUFA-n3 supplementation in this population, particularly among women with a low dietary intake of these fatty acids.

Moreover, even though ART reduces inflammation and immune activation, these levels remain elevated compared to those in healthy individuals, and the imbalance in cytokine profiles persists. ART can also alter cytokine profiles, highlighting the critical need for interventions aimed at reducing chronic inflammation, which can ultimately impact morbidity and mortality in this population.

The relationship between insufficient intake of PUFA-n3 and preterm birth can be attributed to its role in the physiology of delivery. A high ratio of PUFA-n6 to PUFA-n3 may trigger early labor. Therefore, this study aims to evaluate the effects of PUFA-n3 supplementation on birth weight, gestational length, and plasma inflammatory biomarkers in pregnant women using ART.

The sample size for this study was calculated for all the outcome variables. The largest sample size will be used, which was the one calculated to find differences between the means in the IL-6 concentrations of the two supplementation groups, accepting a type I error of 0.05, α=0.05 (1.96), aiming to show a true difference with 0.80 probability, β=0.20 (-0.84). A study in pregnant women was taken as a reference, where the intervention was carried out with a similar dose of PUFA-n3 (1200 mg). The difference found in IL-6 concentrations was 2.8 pg/mL, and following the standard deviation observed in the same study of IL-6 of 4.4 pg/mL. As a result, the sample size will be 38.7 patients per group, plus 20% losses, so 46 patients per group.

The women who meet the inclusion criteria will be invited to participate, and an informed consent letter will be explained and given. Those women who accept will be enrolled in the study. First, they will be randomly assigned to one of the supplementation groups: softgels with 1280mg of PUFA-Ω3 or softgels with a placebo (olive oil).

Allocation to the treatment groups will be done using a table of random numbers, through the software for parallel group clinical trials: Random Allocation Software, created in Microsoft Visual Basic 6 for Windows. Both groups of women will have their usual prenatal care, which includes the Nutrition Care Process. There will be two evaluations, the initial between 20 to 29 weeks of gestational age (GA) according to the first day of the last menstrual period, and the second one, eight weeks after the first (28-37 GA). Both evaluations included: medical history, multiple-pass 24-hour dietary recall, weight measurements, and blood sampling for the inflammatory biomarkers and fatty acid quantification. The pregnancy outcomes, birth weight, and gestational length are going to be obtained from the electronic file. Finally, the statistical analysis will be according to the distribution of outcome variables. The change in the inflammatory biomarkers and the change in the erythrocyte fatty acid profile will be analyzed by a paired t-test or Wilcoxon test. Afterwards, the effect of the supplementation on the pregnancy outcomes and inflammatory biomarkers will be evaluated by the Student t-test or the U-Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Single pregnancy
* Gestational age from 20 to 29 weeks since the first day of the last menstrual period
* Agree to participate in the study

Exclusion Criteria:

* Gestational age more than 29 weeks
* With diagnosis of gestational diabetes or preeclampsia
* Smoking and/or drug use during the invitation to participate in the study
* Fish allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Birth weigth | It will be obtained when the mother's baby is born.
  Birth weight (grams) is the first weight of the fetus or newborn obtained within the first hour of life. It will be obtained from the electronic woman's file.
Length of gestation | It will be obteined and calculated once the mother's baby is born from de electronic file..
  It will be defined as the time (days) between the first day of the mother's last menstrual period and the day of the baby's born.

SECONDARY OUTCOMES:
C-reactive protein (CRP) | It will be obteined from mothers enrollment (20-28 of gestational age) to the end of suplemmentation at 8 weeks.
  C-reactive protein (mg/dL), also called CRP, is a protein made by the liver. The level of CRP increases when there's inflammation in the body. It will be quantified in serum and determined by the immunoturbidimetric method using an analyzer, respons®910 Dyasis brand.
Interleukin 6 (IL-6) | It will be obteined from mothers enrollment (20-28 of gestational age) to the end of suplemmentation at 8 weeks.
  IL-6 (pg/mL) is a soluble mediator with a pleiotropic effect on inflammation, immune response, and hematopoiesis. It will be quantified in serum by an ELISA colorimetric assay using a Benchmark plus reader by Bio-Rad.
Prostaglandin E2 (PGE2) | It will be obteined from mothers enrollment (20-28 of gestational age) to the end of suplemmentation at 8 weeks.
  Prostaglandin E2 (PGE2), a principal mediator of inflammation, plays a critical role in cervical ripening. The quantification will be in serum in pg/mL by an ELISA colorimetric assay using a Benchmark plus reader by Bio-Rad..

OTHER OUTCOMES:
Erythrocyte Fatty Acid Profile | It will be obteined from mothers enrollment (20-28 of gestational age) to the end of suplemmentation at 8 weeks.
  Erythrocyte Fatty Acid (FA) Profile represents the analysis of lipid compositions from mature red blood cell (RBC) membranes in percentage. FA extraction was performed according to Folch's modified method, with an isopropanol-hexane (6.5:4.0) solution. Erythrocytes' FA methyl esters (FAMEs) were separated and measured on a gas chromatograph (Hewlett PackardTM 5890 Series II, Palo Alto, US) coupled to a hydrogen flame detector (FID). It will be the percentage change (% after 8 weeks of supplementation - % basal).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Perinatologia, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Only IPD that will be used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the beginning of the study, and until the end of the study
Access Criteria: Who wanted to know more about this study, and when the results were published, if it is required.

REFERENCES:
- [Background] Valentine CJ, Khan AQ, Brown AR, Sands SA, Defranco EA, Gajewski BJ, Carlson SE, Reber KM, Rogers LK. Higher-Dose DHA Supplementation Modulates Immune Responses in Pregnancy and Is Associated with Decreased Preterm Birth. Nutrients. 2021 Nov 26;13(12):4248. doi: 10.3390/nu13124248. PMID 34959801
- [Background] Best KP, Gomersall J, Makrides M. Prenatal Nutritional Strategies to Reduce the Risk of Preterm Birth. Ann Nutr Metab. 2020;76 Suppl 3:31-39. doi: 10.1159/000509901. Epub 2021 Jan 19. PMID 33465767
- [Background] Nikbakht R, Moghadam EK, Nasirkhani Z. Maternal serum levels of C-reactive protein at early pregnancy to predict fetal growth restriction and preterm delivery: A prospective cohort study. Int J Reprod Biomed. 2020 Mar 29;18(3):157-164. doi: 10.18502/ijrm.v18i3.6710. eCollection 2020 Mar. PMID 32309764
- [Background] Kalagiri RR, Carder T, Choudhury S, Vora N, Ballard AR, Govande V, Drever N, Beeram MR, Uddin MN. Inflammation in Complicated Pregnancy and Its Outcome. Am J Perinatol. 2016 Dec;33(14):1337-1356. doi: 10.1055/s-0036-1582397. Epub 2016 May 9. PMID 27159203
- [Background] Middleton P, Gomersall JC, Gould JF, Shepherd E, Olsen SF, Makrides M. Omega-3 fatty acid addition during pregnancy. Cochrane Database Syst Rev. 2018 Nov 15;11(11):CD003402. doi: 10.1002/14651858.CD003402.pub3. PMID 30480773
- [Background] Serra R, Penailillo R, Monteiro LJ, Monckeberg M, Pena M, Moyano L, Brunner C, Vega G, Choolani M, Illanes SE. Supplementation of Omega 3 during Pregnancy and the Risk of Preterm Birth: A Systematic Review and Meta-Analysis. Nutrients. 2021 May 18;13(5):1704. doi: 10.3390/nu13051704. PMID 34069867
- [Background] Yeganeh N, Watts DH, Xu J, Kerin T, Joao EC, Pilotto JH, Theron G, Gray G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Veloso V, Camarca M, Mofenson L, Moye J, Nielsen-Saines K. Infectious Morbidity, Mortality and Nutrition in HIV-exposed, Uninfected, Formula-fed Infants: Results From the HPTN 040/PACTG 1043 Trial. Pediatr Infect Dis J. 2018 Dec;37(12):1271-1278. doi: 10.1097/INF.0000000000002082. PMID 29750766
- [Background] Shinar S, Agrawal S, Ryu M, Walmsley S, Serghides L, Yudin MH, Murphy KE. Perinatal outcomes in women living with HIV-1 and receiving antiretroviral therapy-a systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2022 Feb;101(2):168-182. doi: 10.1111/aogs.14282. Epub 2021 Oct 27. PMID 34704251
- [Background] Eke AC, Mirochnick M, Lockman S. Antiretroviral Therapy and Adverse Pregnancy Outcomes in People Living with HIV. N Engl J Med. 2023 Jan 26;388(4):344-356. doi: 10.1056/NEJMra2212877. No abstract available. PMID 36720135
- See also: Infectious Morbidity, Mortality and Nutrition in HIV-exposed, Uninfected, Formula-fed Infants: Results from the HPTN 040/PACTG 1043 Trial — https://journals.lww.com/pidj/abstract/2018/12000/infectious_morbidity,_mortality_and_nutrition_in.17.aspx
- See also: Inflammation in Complicated Pregnancy and Its Outcome — https://www.thieme-connect.de/products/ejournals/abstract/10.1055/s-0036-1582397
- See also: Maternal serum levels of C-reactive protein at early pregnancy to predict fetal growth restriction and preterm delivery — https://pmc.ncbi.nlm.nih.gov/articles/PMC7142318/